CLINICAL TRIAL: NCT01848795
Title: Study of Metabolic Effects of EndoBarrier Versus Intragastric Balloon in Obese Patients With Type 2 Diabetes.
Brief Title: EndoBarrier Versus Intragastric Balloon in Obese Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Principal Investigator, Anna Casu, Diabetology Attending, The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRRB/30/10
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 Diabetes; Obesity; gastrointestinal hormones; intestinal bypass; endoscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EndoBarrier Gastrointestinal Liner (Experimental): The treatment in this arm is the endoscopic positioning of the EndoBarrier Gastrointestinal Liner and follow up.
  Interventions: Device: EndoBarrier Gastrointestinal Liner
- Intragastric Balloon (Active Comparator): The treatment in this arm is the endoscopic positioning of the intragastric balloon (Easy life balloon) as a comparator and follow up.
  Interventions: Device: Easy life balloon

INTERVENTIONS:
Device: EndoBarrier Gastrointestinal Liner — Endoscopy placement of EndoBarrier, and clinical and biochemical follow up
  Other Names: produced by GI Dynamics
  Arms: EndoBarrier Gastrointestinal Liner
Device: Easy life balloon — Endoscopy placement of EndoBarrier, and clinical and biochemical follow up
  Arms: Intragastric Balloon

SUMMARY:
Obese patients with Type 2 diabetes (T2D) have a 80-98% chance of having their disease cured or improved following bariatric surgery. This could be explained by weight loss or by changes of nutrient absorption or gut hormone secretion. The comparison of glucose metabolism in patients undergoing malabsorptive or mechanical procedures will clarify this matter. EndoBarrier is an endoscopically delivered device that mimics malabsorptive surgical procedures while the endoscopically placed intragastric balloon induces weight loss with a mechanical action.

The present study hypothesis is that the bypass of the first portion of the intestine obtained with the EndoBarrier will be more effective in improving glucose metabolism than the reduction of food intake obtained with the intragastric balloon. Since similar weight loss is expected in the two groups, the study will aid in understanding the mechanisms behind the metabolic improvement seeing after intestine bypass.

DETAILED DESCRIPTION:
Bariatric surgery is an effective therapy for obesity. Malabsorption-based surgical techniques (excluding the first part of the gastrointestinal tract from the alimentary circuit) are also effective in correcting T2D, even before any significant weight loss has occurred. Proposed mechanisms to explain this beneficial effect include caloric restriction, altered secretion of gut hormones due to duodenal exclusion or due to contact of undigested food with the jejunal mucosa, pancreatic islet hyperfunction, changes of intestinal flora, mucosal inflammation, and/or changes in the biliary acid re-circulation.

EndoBarrier is an endoscopically delivered device that mimics malabsorptive surgical procedures while the endoscopically placed intragastric balloon induces weight loss with a mechanical action.

The present study is a prospective, randomized clinical trial. It will compare the metabolic compensation between patient treated with EndoBarrier and patient treated with Intragastric Balloon.

The aims will be: comparison of glycemic control as measured by hemoglobin A1c (HbA1c), change in oral hypoglycemic drug consumption and body loss from baseline and during follow up in the two groups; evaluation of mechanisms implicated in glycemic control by measuring basal and stimulated insular hormones, glucose levels and gastrointestinal hormones; creation of a bio-bank and dedicated database to collect biological samples for further future studies.

Obese adult T2D patients (BMI ≥ 30) with diabetes duration <10 years will be randomized to receive either EndoBarrier (n=45) or Intragastric Balloon (n=45). The devices will be implanted and kept in place for the first 12 months of study and then removed. Clinical and biochemical data will be collected every 3 months during the 12 months of implant and for the subsequent 12 months after removal.

Statistics describing variables at baseline, at subsequent visits and at the end of the study will be produced for both groups of patients. The Student's t-test will be used for a cross-sectional analysis while the mixed model system will be used for longitudinal observations. Multivariate analysis will also be applied to better characterize differences that may be seen between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-60 year old)
* Type 2 Diabetes diagnosed less than 10 years ago
* Obesity (BMI > 30)

Exclusion Criteria:

* pregnancy
* inflammatory bowel disease
* peptic ulcer
* gastrointestinal disease preventing device positioning
* pancreatitis,
* coronary artery disease
* symptomatic pulmonary disease
* infection at the time of device placement,
* high risk of gastrointestinal bleeding (coagulopathy, bleeding diathesis, anti-coagulant therapy, Non-Steroid Anti-Inflammatory Drugs)
* altered GI anatomy that could affect device placement
* contraindication of positioning of the devices as per technical description of the producer
* C-peptide negative diabetes
* failure to understand the study protocol or not willing to undergo planned follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 12 months
  measurement of diabetes metabolic control

CONTACTS AND LOCATIONS:
Overall Officials: Anna Casu, MD, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- ISMETT, Palermo, Italy, Italy